CLINICAL TRIAL: NCT00787696
Title: HIV Risk Reduction Among Young Incarcerated Females
Brief Title: Healthy Teen Girls: HIV Risk Reduction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mississippi State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Angela A. Robertson, PhD, Research Professor, Mississippi State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA17509-4; R01DA017509 (NIH)
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: HIV-infection/Aids
Keywords: HIV prevention; female adolescent offenders; sexual risk reduction; alcohol and other drug abuse
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Skills Training (Experimental): intervention group received information, motivation and skills training: condom application, assertive communication & problem solving
  Interventions: Behavioral: Cognitive-behavioral HIV/STD risk reduction
- Health Education (Active Comparator): Comparsion group received information and motivation
  Interventions: Behavioral: Cognitive-behavioral HIV/STD risk reduction

INTERVENTIONS:
Behavioral: Cognitive-behavioral HIV/STD risk reduction — 18 60-minute group sessions plus 1 individual health and safety planning session

SUMMARY:
This project assesses the efficacy of an HIV prevention program with adolescent females incarcerated in the Mississippi training school for girls. Participants in both the health education control group and the HIV prevention group will increase health knowledge as a result of their participation in the health classes while incarcerated. However, participants in the HIV prevention group will increase their condom application, assertiveness, and communication skills relative to girls in the health education only group. In addition, after release from the training school, participants in the HIV prevention group will report lower sexual risk behaviors and will have lower rates of infection with chlamydia and gonorrhea during the 12-month follow-up period than participants in the health education only group.

DETAILED DESCRIPTION:
This study is a longitudinal analysis of STD/HIV exposure among adolescent female offenders in Mississippi, a population that is disproportionately African American, and at higher risk than adolescents in general due to their propensity to engage in a variety of risk-taking behaviors, earlier onset of sexual behaviors, and the greater prevalence of mental disorders, substance abuse disorders, maltreatment, and family dysfunction. Based on social cognitive theory and Fisher and Fisher's (1992) IMB (Information, Motivation, and Behavioral skills) model, we will evaluate a drug abuse related HIV risk reduction intervention and compare outcomes against a STD/HIV information and health education control condition.

Approximately 400 females committed to the state reformatory/training school for girls will be recruited for participation. The research design will consist of alternating cohort/waves of about 50 subjects each. One treatment condition will be administered at a time with a washout period between cohort/waves. Over a three year period, one half of subjects will get 18 hours of STD/HIV prevention and one half will get 18 hours of Health Education. All subjects will receive one individual counseling session designed to enhance motivation for behavioral change just prior to release from training school. Before and after the intervention, subjects' social competency skills, condom application skills, and health knowledge will be measured. Before intervention and at 6-month and 12-month follow-up, self-report measures of alcohol and drug use, condom use, sexual risk behaviors, and measures of victimization, partner risk, condom attitudes, self-efficacy, and communication related to condom use and risk reduction will be collected. Urine tests for the detection of 2 STDs (chlamydia and gonorrhea) will also be performed at admission to Columbia Training School and at 6-month and 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Female, ages 13 to 17 years, committed to Columbia Training School, who provide written informed assent.

Exclusion Criteria:

* Acute or chronic physically illness that would preclude participation as determined by facility physician; placement in maximum security unit; study participation during a prior commitment

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 333 (Actual)
Dates: Start 2003-09; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
number of partners and frequency of sexual risk behaviors | at 6 & 12 months
  Sexual behaviors included condom use in the 3 months prior to each assessment. Unprotected sex occasions (USOs) was calculated by subtracting the number of condom-protected vaginal and anal intercourse occasions from the total number of vaginal and anal intercourse occasions. Sex under the influence is the number of times participant reported sexual intercourse after drinking alcohol or using another drug. Safer sex was categorized as sexually abstinent or consistent condom use.
infection with chlamydia or gonorrhea | one year

SECONDARY OUTCOMES:
reproductive health knowledge | pre and post-intervention
  Assessed as the number of correct answers to 37 treu/false and multiple choice questions
condom application skill | pre and post-intervention
  Measured by observing participants apply and remove a condom from a penile model and a 10-item checklist
Communication skills | pre and post-intervention
  Assessed during three role-play vignettes that place the respondent in a high-risk sexual or drug use situation and asked them to respond to a series of three escalating prompts as though the situation was actually happening.
Perceived barriers to condom use | at baseline, 6 and 12 month follow-up
  assessed using the Condom Barrier Scale (St. Lawrence, Chapdeline, et al., 1999)

CONTACTS AND LOCATIONS:
Overall Officials: Angela A. Robertson, Ph.D., Principal Investigator — Mississippi State University
Locations (1):
- Columbia Training School, Columbia, Mississippi, United States

REFERENCES:
- [Result] Robertson AA, St Lawrence J, Morse DT, Baird-Thomas C, Liew H, Gresham K. The Healthy Teen Girls project: comparison of health education and STD risk reduction intervention for incarcerated adolescent females. Health Educ Behav. 2011 Jun;38(3):241-50. doi: 10.1177/1090198110372332. Epub 2011 Mar 10. PMID 21393623